CLINICAL TRIAL: NCT06310122
Title: Effect of Extracorporeal Shockwave Therapy on Gait Parameters in Patients With Plantar Fascitis
Brief Title: Effect of Extracorporeal Shockwave Therapy on Gait Parameters in Patients With Planter Fascitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Elham Mohammed Khairy Abd El Azeem El Naggar, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ESWT on planter fascitis
Record Dates: First submitted 2024-03-04; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Plantar Fascitis; Extracorporeal Shockwave Therapy
MeSH Terms: interventions — Extracorporeal Shockwave Therapy; Ultrasonography

STUDY DESIGN:
Intervention Model Description: Two groups : group (A) , group (B) One of them will receive traditional treatment ( ultra sound , exercises) Other one will recieve extracorporeal shockwave therapy and traditional treatment also
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group (A) treatment group (Experimental): Group (A) will receive extracorporeal shockwave therapy and (Ultrasound, stretching and strengthening exercises)
  Interventions: Device: Extracorporeal shockwave therapy; Device: ultrasound
- Group (B) traditional group (Experimental): Group (B) will receive (Ultrasound, stretching and strengthening exercises)
  Interventions: Device: ultrasound

INTERVENTIONS:
Device: Extracorporeal shockwave therapy — Devices used to improve foot function pain and gait pattern
  Patients will be placed in prone position, therapist locate the point of maximum tenderness. treatment area will be prepared with coupling gel to minimize the loss of shockwave therapy at the interface between applicator tip and skin. Each patient will receive 2000 impulses ,3 bar energy,15mm depth applicator at frequency (10 HZ) per session / week for 4 weeks
  Arms: Group (A) treatment group
Device: ultrasound — Devices used to improve foot function pain and gait pattern
  Participants in the study group will be treated with 5 minutes of therapeutic ultrasound at a frequency of 1 MHz and continuous current at a pulse intensity of 1.8 W/cm2 (when the sensitivity level was too high and the procedure hurt the patient, the therapist reduced the intensity . 3 sessions /week for 4 weeks

SUMMARY:
The purpose of this study is :

* to determine the effect of extracorporeal shockwave on pain intensity in patients with plantar fasciitis.
* to determine the effect of extracorporeal shockwave on foot function in patients with plantar fasciitis.
* to determine the effect of extracorporeal shockwave on gait parameters in patients with plantar fasciitis

DETAILED DESCRIPTION:
Plantar fasciitis with an accompanying heel spur is very burdensome and difficult to treat disease. It most often arises as a result of degenerative changes of the proximal plantar fascia and the tissues surrounding the aponeurosis, occurring due to continuous irritation of the area and resulting micro-injuries. The main symptom of plantar fasciitis is pain in the heel area; this worsens over time, increasingly occurring upon loading and eventually, even at rest. Redness and swelling are also observed in the heel. The risk of the disease is increased by being overweight, working a job that requires long periods of standing, lifting heavy objects.

About 85% to 90% of patients do not need to undergo surgery, and 80% of patient do not experience pain relapse after conservative treatments. Minimally invasive treatments commonly used for treating PF are extracorporeal shockwave therapy (ESWT), corticosteroid (CS)injections, platelet-rich plasma (PRP) injections, botulinum toxin (BTX), acupuncture, dry needling and prolotherapy.

Conservative treatment options for PF include rest, weight loss, non-steroidal anti-inflammatory drugs, physical therapies (ultrasound therapy, low-energy, and laser therapy), plantar fascia and calf muscle strengthening and stretching exercises. If symptoms persist, second-option treatment is usually local corticosteroid injections. However, despite providing a good effect in terms of pain reduction, corticosteroids have proven to damage the fascial tissue, thus increasing the risk of further degeneration and eventual rupture. To avoid this complication, Extracorporeal shock wave therapy (ESWT) is a treatment recommendation for patients with chronic PF recalcitrant to other conservative treatment.

Extracorporeal shockwave therapy (ESWT) is a physical therapy that generates three-dimensional pressure pulses, lasting microseconds and reaching peek pressures of 35-120 MPa, and has effects depending on intensity, pulse cycle and shockwave (SW) modality. We have two modalities of SW therapy: focused shockwave (FSW) and radial shockwave (RSW). FSW is documented as a possible alternative to the surgical approach: it focuses on a small area (2 to 8 mm) and penetrates at a selected depth, having effects that depend on the energy delivered to the focal area; that is why it is important to know the energy flux density (EFD), which is considered the "dose" of SW administered.

RSW produces SW that are transmitted radially and do not have penetrating effects on tissue, acting superficially. They are frequently used in soft-tissue pathologies and, recently, also in plantar fasciitis. As this physical therapy is widely used for the treatment of plantar fasciitis. The mechanism of ESWT is not completely clear. However, it is speculated that ESWT may produce a reflexive analgesic effect by inducing excitability of the axon and destroying unmyelinated sensory fibers.

Due to the negligible side effects, which only relate to minor referred pain during ESWT sessions and minor hematoma, this therapy represents a safe, advantageous, and well-tolerated approach without surgical risks or severe complications. Therefore, the use of ESWT has gained increasing popularity for treating different musculoskeletal disorders. These encompass tendinopathies (both calcifying and non-calcifying), plantar fasciitis (PF), lateral epicondylitis ("tennis elbow"), greater trochanteric pain syndrome, bone nonunion fractures, and joint diseases including avascular necrosis.

The extracorporeal shock wave produces a treatment effect by passing through muscle and adipose tissue and releasing energy at the border of the bone due to the difference in impedance. Therefore, ESWT improves the clinical condition of the plantar fascia. Thus, the benefits of ESWT may be fundamentally more difficult to achieve in patients with pain throughout the entire plantar fascia when the ESWT target site is far from the enthesis of the calcaneus. Furthermore, the investigators speculate that the ESWT effect may be insufficient in patients with degeneration of the plantar fascia itself.

ELIGIBILITY:
Inclusion Criteria:

* - 52 female patient with chronic planter fasciitis.
* Patient,s age will be (18 - 40) , all of them are diagnosed with planter fasciitis will be recruited for the study.
* BMI will be (18 - 40 kg/m2).
* Unilateral chronic planter fasciitis.
* Symptoms of pf pain lasted more than 3 months.
* Diagnosis of painful heel syndrome by clinical examination, with the following positive clinical signs:

  * Pain in the morning or after sitting a long time.
  * Local pain where the fascia attaches to the heel.
  * Increasing pain with extended walking or standing for more than 15 minutes.
  * History of 6 months of unsuccessful conservative treatment.
* Therapy free period of at least 4 weeks before referral.

Exclusion Criteria:

Patients will exclude from this study if their pain due to:

* Bilateral plantar fasciitis.
* Dysfunction of foot or ankle (for example, instability).
* Arthrosis or arthritis of the foot.
* Infections or tumors of the lower extremity.
* Neurological abnormalities, nerve entrapment (for example, tarsal tunnel syndrome).
* Vascular abnormality (for example, severe varicosities, chronic ischemia).
* Operative treatment of the heel spur.
* Hemorrhagic disorders and anticoagulant therapy.
* Pregnancy.
* Diabetes.
* Trauma.
* previous surgery.
* Inflammation disease.
* Rheumatoid arthritis

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-03-12 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Stride length mean distance measured by (meter) | 4 weeks
  stride length (one of gait parameters) that will be assessed by using Kinovea software.
stride time mean time measured by (second) | 4 weeks
  stride time (other gait parameters) that will be assessed by using kinovea software
speed mean distance/ time measured by (meter/second) | 4 weeks
  speed (other gait parameters) that will be assessed by using kinovea software.
cadence mean number of steps /times. | 4 weeks
  cadence (other gait parameters) that will be assessed by using kionvea software.

SECONDARY OUTCOMES:
pain intensity level. | 4 weeks
  pain intensity will be assessed by visual analogue scale. 0 mean (no pain) that mean better outcomes to 10 that mean (unbearable pain) that mean worst outcomes.

OTHER OUTCOMES:
Foot function | 4 weeks
  foot function will be assessed by foot function index. 0 mean (no pain or difficulty) that mean better outcomes to 10 (worst pain imaginable or so difficult it requires help) that mean worst outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Amir M Saleh, Professor, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Latt LD, Jaffe DE, Tang Y, Taljanovic MS. Evaluation and Treatment of Chronic Plantar Fasciitis. Foot Ankle Orthop. 2020 Feb 13;5(1):2473011419896763. doi: 10.1177/2473011419896763. eCollection 2020 Jan. PMID 35097359
- [Background] Greve JM, Grecco MV, Santos-Silva PR. Comparison of radial shockwaves and conventional physiotherapy for treating plantar fasciitis. Clinics (Sao Paulo). 2009;64(2):97-103. doi: 10.1590/s1807-59322009000200006. PMID 19219314
- [Background] Lai TW, Ma HL, Lee MS, Chen PM, Ku MC. Ultrasonography and clinical outcome comparison of extracorporeal shock wave therapy and corticosteroid injections for chronic plantar fasciitis: A randomized controlled trial. J Musculoskelet Neuronal Interact. 2018 Mar 1;18(1):47-54. PMID 29504578